CLINICAL TRIAL: NCT03512873
Title: A Clinical Study of Tranilast in the Treatment of Scleredema Diabeticorum
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH Hou
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-01

CONDITIONS: Scleredema Adultorum
Keywords: Scleredema Diabeticorum; Tranilast
MeSH Terms: conditions — Scleredema Adultorum | interventions — tranilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tranilast (Experimental)
  Interventions: Drug: Tranilast

INTERVENTIONS:
Drug: Tranilast — Subjects will be treated with tranilast

SUMMARY:
56 patients with scleredema diabeticorum will be selected to receive treatment of tranilast. After a period of time ,we can determine the efficacy of the drug by detecting the the thickness of skin before and after treatment.

DETAILED DESCRIPTION:
56 patients with Scleredema Diabeticorum will be selected. After the signing of the informed consent ,they will be collected the initial lesions photos,the thickness of skin lesions by ultrasound and magnetic resonance,and chemical examinations including blood routine examination, routine urine test, liver function, renal function.During tranilast (0.1g each time, three times a day,6 months) treatment, patients need regular follow-up (1 per month) including liver and kidney function, blood glucose level monitoring, and every three months to retest lesion thickness.With 3 month as a time point, they were observed for two points.After the experiment, the experimental data will be arranged and the data of the thickness change of skin lesions will be statistically processed (t test) to determine whether it is meaningful.

ELIGIBILITY:
Inclusion Criteria:

* (1)Clinical and histopathological examination has been proved to be scleredema diabeticorum; (2)Ultrasound and magnetic resonance detection found that the thickest skin of the back was more than 5mm.

Exclusion Criteria:

* (1)with a liver or kidney disease, or accompanied by a tumor or a severe infection ; (2)Poor blood sugar control; (3)with mental disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Measure the volume change of skin lesions by ultrasound | This experiment will last for 6 months
  During tranilast (0.1g each time, three times a day, 6 months) treatment, patients need to test lesion volume.The reduction of volume greater than 50% is judged to be effective